CLINICAL TRIAL: NCT01686620
Title: A Randomized, Parallel Group Trial Evaluating Safety and Efficacy of BIOD-123 Compared to Insulin Lispro (Humalog®) in Subjects With Type 1 Diabetes Using Basal-bolus Insulin Injection Therapy
Brief Title: A Study Evaluating Safety and Efficacy of BIOD-123 Compared to Insulin Lispro (Humalog®)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-201
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Mealtime insulin; Ultra-rapid acting insulin; Prandial insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIOD-123 (Experimental): BIOD-123 used as prandial insulin
  Interventions: Drug: BIOD-123
- Lispro (Humalog) (Active Comparator): Lispro (Humalog) used as prandial insulin
  Interventions: Drug: Lispro (Humalog)

INTERVENTIONS:
Drug: BIOD-123
  Arms: BIOD-123
Drug: Lispro (Humalog)
  Arms: Lispro (Humalog)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BIOD-123 compared to insulin lispro (Humalog®) when used as part of a basal-bolus regimen in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of type 1 diabetes, consistent with ADA classification criteria (Diabetes Care 35: S64-S71, 2012), for more than 1 year.
* Age: 18 years old, or older.
* Body Mass Index: between 18 and 35 kg/m2, inclusive.
* Willing to use insulin glargine as the only basal insulin throughout the duration of the trial.
* Willingness not to use insulin pump treatment and only use the study glucose meter and CGM devices during the duration of the trial.

Exclusion Criteria:

* History of known hypersensitivity to any of the components in the study medication
* Treatment with pramlintide or GLP-1 analogs within 30 days of screening or anticipated use of these medications during the course of the study.
* Treatment with oral or intravenous corticosteroids in the last 3 months prior to screening. Standard doses of inhalational corticosteroid used as part of a long term treatment regimen are allowed.
* Consistent recent hypoglycemic unawareness within the last six months
* History of more than two severe hypoglycemic events within six months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C | Baseline and 18 week treatment period

SECONDARY OUTCOMES:
Hypoglycemic event rates | Baseline and 18 week treatment period
Insulin dose | Baseline and 18 week treatment period
Daily blood glucose measures | Baseline and 18 week treatment period

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Profil Research Institute, Chula Vista, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Private Practice - Richard Cherlin, MD., Los Gatos, California
  - Providence Clinical Research Pharmaseek, North Hollywood, California
  - Monteagle Medical Center, San Francisco, California
  - Mills-Peninsula Health Services, San Mateo, California
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - University of Miami Diabetes Research Institute, Miami, Florida
  - Progressive Medical Research Pharmaseek, Port Orange, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center PA, Idaho Falls, Idaho
  - MidAmerica Diabetes Associates, PA, Wichita, Kansas
  - Kentucky Diabetes, Lexington, Kentucky
  - Diabetes & Glandular Disease Research, Rockville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mercury Street Medical, Butte, Montana
  - Desert Endocrinolgy, Henderson, Nevada
  - Research Foundation of SUNY Upstate Medical University, Syracuse, New York
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Sentral Clinical Research Services, LLC, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Mountain Diabetes & Endrocrine Center, Dallas, Texas
  - Dallas Diabetes and Endocrine Research Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Sonterra Clinical Research, San Antonio, Texas
  - Capital Clinical Research Center, Olympia, Washington
  - Ranier Clinical Research, Inc, Renton, Washington
  - Rockwood Clinic, Spokane, Washington